CLINICAL TRIAL: NCT06378333
Title: Incidence, Clinical Characteristics and Outcomes of Unstable Angina in the contempoRary Area. ICAR Observational Study
Brief Title: Incidence, Clinical Characteristics and Outcomes of Unstable Angina in the contempoRary Area.
Acronym: ICAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01-023
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Unstable Angina
Keywords: cardiology
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: patients who underwent coronary angiography — All patients included in the ICAR project (Montpellier - Nîmes) benefit from a consultation at one year (12+or - 2 months), as they are systematically reviewed in our department: data will therefore be collected in the patient's medical record. Clinical biological parameters and events during the hospital phase are also collected in the patient's computerized record. Normal patient management remains unchanged.

SUMMARY:
The study aims to evaluate clinical characteristics and prognostic of a contemporary population of patients with UA defined using T hs-cTn measurements The study includes all patients admitted in 2 French university centers with the confirmed diagnostic of UA defined with clinical ischemic symptoms and T hs-cTn concentrations < 99 percentile (undetectable: <5ng/l or non-elevated: <14ng/l), or ≥ 99 percentile but mildly elevated (14-50ng/l) .The primary end-point included major events at 1-year follow-up (total mortality, new ACS, hospitalization for cardiac causes).

ELIGIBILITY:
Inclusion criteria:

* Patients with ischemic symptoms at rest or minor exercise without evidence of acute myocardial necrosis.
* Ischemic symptoms may include typical or atypical angina pectoris and worsening/deterioration of previously stable angina with or without electrical signs of ischemia on the electrocardiogram.
* hs-cTn concentrations are in the normal range or may be slightly elevated > 99th percentile (i.e. low troponin T elevation ≤ 50 * Elecsys Roche) but with absence of significant kinetics according to criteria defined in the literature (<20%).
* One of the following angiographic criteria is required:

  * Coronary angiography revealing a stenosis with a diameter of at least 70%.
  * Stenosis of at least 50% diameter in the left common trunk.
  * FFR (Fractional Flow Reserve) documenting ischemia per coronary angiography of a coronary lesion in the case of intermediate stenosis (50-70%).
  * If there are no significant lesions, a spasm must be proven by an ergonovine test.

Exclusion criteria:

* NSTEMI and STEMI.
* Coronaries normal or without significant lesions unless proven spasm.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unstable angina proven by coronary angiography admitted to Montpellier and Nîmes hospitals between November 2021 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with hospitalisation for unstable angina | One year after hospitalisation for of unstable Angina

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PUPH, Study Director — Montpellier University Hospital
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamm CW, Braunwald E. A classification of unstable angina revisited. Circulation. 2000 Jul 4;102(1):118-22. doi: 10.1161/01.cir.102.1.118. PMID 10880424
- [Background] Puelacher C, Gugala M, Adamson PD, Shah A, Chapman AR, Anand A, Sabti Z, Boeddinghaus J, Nestelberger T, Twerenbold R, Wildi K, Badertscher P, Rubini Gimenez M, Shrestha S, Sazgary L, Mueller D, Schumacher L, Kozhuharov N, Flores D, du Fay de Lavallaz J, Miro O, Martin-Sanchez FJ, Morawiec B, Fahrni G, Osswald S, Reichlin T, Mills NL, Mueller C. Incidence and outcomes of unstable angina compared with non-ST-elevation myocardial infarction. Heart. 2019 Sep;105(18):1423-1431. doi: 10.1136/heartjnl-2018-314305. Epub 2019 Apr 24. PMID 31018955
- [Background] Kristensen AMD, Pareek M, Kragholm KH, Sehested TSG, Olsen MH, Prescott EB. Unstable Angina as a Component of Primary Composite Endpoints in Clinical Cardiovascular Trials: Pros and Cons. Cardiology. 2022;147(3):235-247. doi: 10.1159/000524948. Epub 2022 May 10. PMID 35537418
- [Background] Eggers KM, Jernberg T, Lindahl B. Unstable Angina in the Era of Cardiac Troponin Assays with Improved Sensitivity-A Clinical Dilemma. Am J Med. 2017 Dec;130(12):1423-1430.e5. doi: 10.1016/j.amjmed.2017.05.037. Epub 2017 Jun 21. PMID 28647406
- [Background] Vafaie M, Slagman A, Mockel M, Hamm C, Huber K, Muller C, Vollert JO, Blankenberg S, Katus HA, Liebetrau C, Giannitsis E, Searle J. Prognostic Value of Undetectable hs Troponin T in Suspected Acute Coronary Syndrome. Am J Med. 2016 Mar;129(3):274-82.e2. doi: 10.1016/j.amjmed.2015.10.016. Epub 2015 Oct 30. PMID 26524709
- [Background] Olivier CB, Sundaram V, Bhatt DL, Leonardi S, Lopes RD, Ding VY, Yang L, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, White HD, Desai M, Lynch DR Jr, Harrington RA, Mahaffey KW; CHAMPION PLATFORM and CHAMPION PCI Investigators. Definitions of peri-procedural myocardial infarction and the association with one-year mortality: Insights from CHAMPION trials. Int J Cardiol. 2018 Nov 1;270:96-101. doi: 10.1016/j.ijcard.2018.06.034. Epub 2018 Jun 8. PMID 29937301
- [Derived] Jouen R, Meunier PA, Moulis L, Roubille F, Macia JC, Berdeu JM, Steinecker M, Robert P, Lattuca B, Cayla G, Leclercq F. Incidence and 1-Year Prognostic of Unstable Angina After High-Sensitivity Troponin Assessment. Catheter Cardiovasc Interv. 2025 May;105(6):1445-1452. doi: 10.1002/ccd.31473. Epub 2025 Mar 6. PMID 40047210